CLINICAL TRIAL: NCT06605573
Title: Lay User Evaluation of the Panbio™ HCV Self Test: a Prospective, Multi-centre Observed Untrained User Study.
Brief Title: Lay User Evaluation of the Panbio™ HCV Self-Test
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Rapid Dx (Industry)
Collaborators: Aga Khan University (Other); Clinic 553 Karachi (Unknown); Ezintsha Clinical Research Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: SDRD-I-030-P
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: HEPATITIS C (HCV)
Keywords: diagnostics; rapid test; untrained user; hepatitis C; lateral flow test
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: Single group assessment
Who Masked: Outcomes Assessor
Masking Description: The study staff member who interprets the lay user's result will be blinded to the lay user's reference test results and medical status. The study staff member who conducts the Panbio™ HCV Self Test for the lay user will also be blinded to the lay user's reference test results and medical status as well as the self-test results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Panbio™ HCV Self Test — Rapid diagnostic test (self-test and professional) plus laboratory reference tests
  Other Names: Fingerstick HIV testing (optional); Laboratory reference testing for HCV (immunoassays and PCR, CE marked)

SUMMARY:
This is a prospective, multi-centre study designed to evaluate the usability of the Panbio™ HCV Self Test, when performed by untrained lay users in an observed study setting. The Panbio™ HCV Self Test detects antibodies to Hepatitis C Virus (HCV). The study validation will be conducted in accordance with the World Health Organisation's technical guidance on Hepatitis C rapid diagnostic tests for professional use and/or self-testing (TSS-16).

DETAILED DESCRIPTION:
Hepatitis C is a liver disease caused by the hepatitis C virus. The virus can cause both acute and chronic disease, ranging in severity from a mild illness lasting a few weeks to a serious, lifelong illness. Globally, Hepatitis C virus infects around 71 million people per year, resulting in 700,000 deaths. The WHO estimates that only 21% of individuals chronically infected with HCV are diagnosed, and the WHO HCV targets include increasing the diagnoses to 90% by 2030. WHO guidelines, published in 2021, strongly recommend offering self-testing for HCV as an additional approach to HCV testing services.

ELIGIBILITY:
Inclusion Criteria:

* Participant is aged 14 or over
* Participant agrees to all aspects of the study and is able and willing to provide informed consent / assent with parental consent.

Exclusion Criteria:

* Participant has already participated in this study on a previous occasion.
* Participant is aware of their HCV status
* Participant is deemed unfit for the study by the Investigator.
* Participant has a condition deemed unfit by the Investigator to safely perform or receive the test.
* Participant is a practising health-care professional or laboratory scientist / technician or has prior medical or laboratory training or experience
* Participant is currently enrolled in a study to evaluate an investigational drug or vaccine.
* Participant has a visual impairment that cannot be restored using glasses or contact lenses or is unable to read the Instructions for Use.
* Participant is unwilling or unable to provide informed consent.
* Participant has participated in the study "Lay user evaluation of the Panbio™ HCV Self Test: A prospective, multi-centre usability study to evaluate lay user labelling comprehension and test result interpretation".

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1185 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Lay user / professional user test result concordance | 5 months
  To assess the concordance between the Panbio™ HCV Self Test, as performed by lay users based on self-collected finger-stick samples, and the Panbio™ HCV Self Test performed by a trained health care worker, who also will collect the finger-stick sample required for the test and perform the test.
Lay user / laboratory test result concordance | 5 months
  To establish clinical performance (concordance with the reference test) for the Panbio™ HCV Self Test, as performed by lay users using finger-stick whole blood samples, when compared to reference testing using venous plasma samples.

SECONDARY OUTCOMES:
Usability evaluation - lay user experience | 5 months
  To assess the usability of the Panbio™ HCV Self Test, as performed by lay users, based on a participant questionnaire evaluation by the lay user participant. The participant questionnaire includes questions to assess the lay users' experience when performing the test. Most questions have a Yes / No answer option, with free text possible. Some questions require a free text answer.
Usability evaluation - Self-test observer records | 5 months
  To assess the usability of the Panbio™ HCV Self Test, as performed by lay users based on a questionnaire evaluation by the study staff observer. In the observer questionnaire, particular attention will be paid to compliance regarding factors considered critical for the test, such as reading the IFU/ QRG and applying the correct test volume. The observer questionnaire is not reporting scores on a scale, but is recording observations regarding how the users complete each step. For each step, a question is asked whether the user conducted a certain procedure, and a Yes / No answer is requested, with Monitor Notes when applicable.
Lay user / professional user results interpretation concordance | 5 months
  To assess the concordance between the self-test results (obtained by the self-tester) when interpreted by the lay user and by the observer.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Qureshi, MD, Principal Investigator — Clinic 553; Saeed Hamid, Pr, Principal Investigator — Aga Khan University; Mohammed Majam, BSc, MBA, Principal Investigator — Ezintsha

IPD SHARING:
Plan to Share IPD: No